CLINICAL TRIAL: NCT06417164
Title: Effects of FMS Functional Movement Training on Body Posture Control in College Female Aerobics Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lan Li (Other)
Responsible Party: Sponsor-Investigator, Lan Li, lecturers, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LLi
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Postural Balance
Keywords: Posture control; Functional movement training; Randomized controlled trial,

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: 1. Participants do not know which group they have been assigned to (treatment or control). This can be done by providing all participants with the same information after grouping, without revealing which group they are in, to ensure that they do not know which intervention they are receiving.
  2. Trainer blinding is when the trainer does not know which group the participant is in. This can be done by assigning participants to groups by another researcher or by a randomization system to avoid the trainer knowing the participant's group.
  3. Outcome assessment is performed by a researcher who does not know the group the participant is in, hiding information about the participant's group, and using a researcher who is independent of the intervention assignment to perform the outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, Traditional Physical Training Group (No Intervention): The control group will use traditional physical training methods.
- Intervention, Functional Training Group, (Experimental): Intervention, Functional Training Group will use functional movement training methods based on FMS.
  Interventions: Behavioral: Functional Movement Training Group

INTERVENTIONS:
Behavioral: Functional Movement Training Group — The program control group will use traditional physical training methods, while the experimental group will use a training program based on FMS functional movement design. The experimental group will receive a 12-week FMS functional movement training intervention, with each session lasting 40 minutes. The experimental group will be divided into two phases, a corrective intervention phase and a capacity enhancement phase, and the main assessment criteria will include the seven movements of the FMS Functional Movement Test (squat, hurdle step, deep squat, shoulder mobility, active straight leg raise, trunk stabilizing push-ups, and trunk rotational stabilization), as well as the ability to control the body's dynamic and static postures during aerobic exercise.
  Arms: Intervention, Functional Training Group,

SUMMARY:
For this experiment, it was planned to randomly assign 40 female college aerobics athletes to two groups: a traditional physical training group (control group, T, N=20) and a functional training group (experimental group, F, N=20). The control group will use traditional physical training methods, while the experimental group will use a training program based on the FMS functional movement design. The experimental group was scheduled to undergo a 12-week FMS functional movement training intervention, with each session lasting 40 minutes. Before and after the experiment, the subjects' FMS scores, body posture control, and competition performance will be measured.

DETAILED DESCRIPTION:
Randomized into: Control, Traditional physical training Group, T, N = 20 , Intervention, Functional training Group, F, N = 20). The control group used traditional physical training methods, and the experimental group used FMS-based functional movement training methods. A 12-week functional movement training program was used and the experimental group was given intervention training 4 times a week for 40 min each time, and FMS scores, body posture control, and athletic performance were tested before and after the intervention. It was expected that the main assessment criteria would include the seven movements of the FMS Functional Movement Test (deep squat, hurdle step, lunge squat, shoulder flexibility, active straight leg raise, trunk stability push-up, and trunk rotational stability) as well as dynamic and static body postural control in aerobics movements. Tests of T-run and basic pace Y-jump time and athletic performance were used as secondary outcomes. The main tools included: a set of FMS tester, a roll of yellow tape, a measuring tape, a stopwatch, and a test chart for each index.

The test was divided into two phases. Phase 1: corrective training (1-4 weeks), Phase 2 is: the overall movement (functional patterning) 5-12 weeks, while the design concept of the program is shown in the increase of difficulty, specialization, but also includes the process of static stability to dynamic stability, and then finally, the overall movement pattern training. Tools used: balance disk, Swiss ball, solid ball, foam shaft, massage stick.

ELIGIBILITY:
Inclusion Criteria:

① Must be able to understand and comply with the study regulations and sign an informed consent form.

② Have a stable summer training schedule with no plans to return home during the summer.

③ No serious diseases or complications.

Exclusion Criteria:

Athletes with recent sports injuries who may not participate in the training program.

Ages: 18 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-25 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
FMS Score | 90days
  FMS test scores( in points)
Eight-stage abdominal bridge | 90days
  Control of body posture stability under static conditions, ( in points)
five-step lateral bridge | 90days
  Control of frontal body posture stability under static conditions (in points)
six supine bridge | 90days
  Control of back and hip stability under static conditions (in points)

SECONDARY OUTCOMES:
T-type running | 90days
  examine the control ability of the unilateral lower limb of the aerobic athlete's body posture in the rapid and dynamic state.（second ）
Y-type jumping | 90days
  The body posture control test under the conditions of dynamic movement surface change（second ）
Aerobics competitive performance | 90days
  Four groups of difficulty combinations ABCD and single competition routines were used for comprehensive scoring（points）

CONTACTS AND LOCATIONS:
Overall Officials: Zijian Zhao, Study Chair — Zhengzhou University
Locations (1):
- ZhengZhouU, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Yes
All IPDs collected, all IPDs used as a basis for results in publications.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: October 2024